CLINICAL TRIAL: NCT01599533
Title: Screening for Thoracic Aortic Aneurysm Among a Cohort of Patients With a Degenerative Abdominal Aortic Aneurysm : Prevalence, Description of the Different Thoracic Aortic Phenotypes by Aortic Volumetric Numerized Imaging and Their Relationship With Epidemiologic, Clinical, Biological and Genetic Factors
Brief Title: Screening for Thoracic Aortic Aneurysm Among a Cohort of Patients With a Degenerative Abdominal Aortic Aneurysm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-A00042-41; 2012-01 (Other: AP HM)
Record Dates: First submitted 2012-04-10; First posted 2012-05-16 (Estimated); Last update posted 2019-12-02 (Actual); Status verified 2019-10

CONDITIONS: Abdominal Aortic Aneurysms
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- abdominal aortic aneurysms (Other)
  Interventions: Other: blood samples

INTERVENTIONS:
Other: blood samples

SUMMARY:
Many publications deal with the natural history of aortic aneurysms in literature. Except for connective tissue disorders as Marfan or Loeys-Dietz syndrome, aortic aneurysms are a complex multifactorial disease with genetic and environmental risk factors. Susceptibility loci identified in thoracic aortic aneurysms (TAA) and abdominal aortic aneurysms (AAA) do not overlap, suggesting that different genetic risk factors contribute to these two forms of aneuryms. With a higher prevalence correlated to ageing (5%), AAA is usually presented as the degenerative form of the disease. However, a recent epidemiologic study by Olsson et al. has revealed an increasing incidence of thoracic aortic disease among older individuals (70+/-12 years) with 60% of aneurysmal rupture or dissection at diagnosis, and a 1.7 :1 male-to-female ratio compared to 6:1 in AAA. From this current knowledge arises the concept of diffuse or plurisegmental degenerative aneurysmal aortic disease, poorly explored so far. As regards to the prevention policy, there is a consensus statement in which ultrasonography screening for AAA is recommended for all individuals aged > 60 years (particularly in men who have ever smoked) and for those aged > 50 years with family history of AAA. Nevertheless, screening for a concomittant thoracic location of the disease (except thoracoabdominal aneurysm) is not yet required, whereas it could change the prognosis of the patients and influence their management.

DETAILED DESCRIPTION:
Through the constitution of a multicentric prospective cohort of patients with infra-renal AAA (n=450), the investigators aimed to determine the prevalence of a concomitant TAA, and the epidemiologic, clinical, biological and genetic factors related to this aortic phenotype. Therefore, the investigators postulate for a prevalence of the AAA-TAA association inferior or equal to 15%. By the use of an innovating software (AMIRA) to analyse scans, the investigators will perform reproductive measurements of segmental diameters from a segmental aortic volumetric numerized imaging, and describe the different thoracic aortic phenotypes associated with AAA, including the form (TAA, penetrating ulcer, dolichoaorta …) and the location of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Major subject at the time of the inclusion
* Subject sent in hospitalization or in consultation of surgery vascular for coverage of the first one anévrysme of the sub-renal abdominal aorta degenerative, without anomaly associated by the coeliac aorta, and by the upper diameter in 40mm (according to the criteria of measure recommended for the analysis in echography doppler or in angioscanner).
* subject not presenting contraindication to the realization of the diagnostic examination by aortic angioscanner
* Subject having signed a consent.

Exclusion Criteria:

Subject under age 18

* pregnant Woman
* Subject received in the phase aigue of a break or a fissuring of an AAA under renal
* Subject already operated for a thoracic or abdominal aortic anévrysme
* Subject presenting at least one of the following pathologies:
* heart disorder valvulaire aortic: aortic incapacity of rank superior to 2, tight aortic stenosis, prosthesis valvulaire aortic
* context of bicuspidie station wagon diagnosed on at least 2 parents of the first degree
* of a not degenerative aortopathie anévrysmale bound(connected) in bicuspidie aortic, or: A dissection of type(chap) A or of type(chap) B
* Of a degenerative aortopathie of type anévrysme thoracoabdominal (in particular, affected by the coeliac aorta, defined by the segment enter the diaphragmatique crossing and the renal arteries)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
BLOOD SAMPLES | 3 YEARS
  to determine the prevalence thoracic aortic aneurysms (TAA) and abdominal aortic aneurysms (AAA)

SECONDARY OUTCOMES:
ANGIOSCAN | 3 YEARS
  the validation of volumetric criteria to quantify the aortic remodeling in TAA or untreated AAA
CARDIAC STATEMENT | 3 YEARS
  cardiac echography

CONTACTS AND LOCATIONS:
Overall Officials: BERNARD BELAIGUES, Study Director — Assistance Publique hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France